CLINICAL TRIAL: NCT01477372
Title: Effect of Physical Exercise Program During Pregnancy on Excessive Weight Gain and Its Consequences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Politecnica de Madrid (Other)
Responsible Party: Principal Investigator, Ruben Barakat Carballo, Director, Universidad Politecnica de Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 240/09
Record Dates: First submitted 2011-09-22; First posted 2011-11-22 (Estimated); Last update posted 2012-04-11 (Estimated); Status verified 2012-04

CONDITIONS: Pregnancy
Keywords: Pregnancy; Exercise; Excessive weight gain; Outcomes; Urinary incontinence
MeSH Terms: conditions — Motor Activity; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): Supervised exercise program
  Interventions: Behavioral: Supervised exercise program
- Control (No Intervention): Sedentary pregnant woman

INTERVENTIONS:
Behavioral: Supervised exercise program — Intervention group participated in Blooming Exercise Program as from week 10-12 of gestation. At least 56 sessions through 22 weeks. 3 sessions per week
  Arms: Exercise group

SUMMARY:
The purpose of this study was to assess the effectiveness of a moderated physical exercise program called Blooming Exercise Program (BEP) developed during pregnancy in order to control excessive maternal weight gain and its consequences. Additionally, other objectives of the study were to analyse the influence of BEP on urinary incontinence, on the other pregnancy outcomes and on the perception of the pregnant's health

DETAILED DESCRIPTION:
BACKROUND: Pregnancy and delivery can condition significantly women's health. In particular, an excessive gain of weight during pregnancy constitutes a risk factor which may lead to (i) different alterations during pregnancy such as gestational diabetes or hypertension, (ii) foetus health problems (macrosomia), (iii) delivery complications (dystocia, prolonged labour and increased number of caesareans) and (iv) future health disorders for the woman (overweight, obesity and cardiovascular alterations). Furthermore, during pregnancy pelvic floor health problems, such as urinary incontinence (IU) may arise or worsen.

OBJECTIVES: The main aim of this study was to assess the effectiveness of a moderate physical exercise program called Blooming Exercise Program (BEP) developed during pregnancy in order to control excessive maternal weight gain and its consequences. Additionally, other objectives of the study were to analyse the influence of BEP on urinary incontinence, on the other pregnancy outcomes (maternal and foetal) and on the perception of the pregnant's health.

DESIGN: A randomized, controlled trial called has been conducted. 300 healthy pregnant women were recruited and divided into an intervention group (IG, n=100) and a control group (CG, n=200). The IG participated in BEP as from week 10-12 of gestation (at least 56 sessions through 22 weeks. 3 sessions per week). The CG did not participate in any supervised program addressed to pregnant women but received regular health care. Pregnancy outcomes regarding the mother and the new born, urinary incontinence and women's habits data were obtained and registered through initial interviews, medical records and two specific questionnaires on health and urinary incontinency (ICIQ-SF and King's).

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnant women
* Delivering in "Hospital Universitario de Fuenlabrada"
* At week 10-14 of gestation
* Able to attend 3 sessions per week until the end of the pregnancy

Exclusion Criteria:

* Contraindications appointed by ACOG
* Less than 56 sessions

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2007-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Maternal weight gain | week 36-38 of gestation
  Maternal weight gain and proportion of participants exceeding weight gain above IOM (2009) recommendations

SECONDARY OUTCOMES:
Excessive weight gain related risks (gestational diabetes, macrosomia, type of delivery) | week 36-38 of gestation
Urinary incontinence | week 36-38 of gestation
Other pregnancy outcomes (maternal and foetal) | week 36-38 of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Ruben O Barakat, PhD, Study Director — Universidad Politecnica de Madrid; Mireia Peláez, PhD, Principal Investigator — Universidad Politecnica de Madrid
Locations (1):
- Universitarian Hospital of Fuenlabrada, Fuenlabrada, Madrid, Spain

REFERENCES:
- [Derived] Pelaez M, Gonzalez-Cerron S, Montejo R, Barakat R. Protective Effect of Exercise in Pregnant Women Including Those Who Exceed Weight Gain Recommendations: A Randomized Controlled Trial. Mayo Clin Proc. 2019 Oct;94(10):1951-1959. doi: 10.1016/j.mayocp.2019.01.050. PMID 31585579